CLINICAL TRIAL: NCT06839625
Title: The Effect of Emotional FreedomTechnique on Postoperative Pain, Pain Belief and Anxiety in Coronary Artery Bypass Graft Planned Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Collaborators: Samsun Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Özge İşeri, Assistant Professor, Ondokuz Mayıs University, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-26521195-604.01-262284337; Ondokuz Mayıs University (Other: Ondokuz Mayıs University)
Record Dates: First submitted 2025-02-12; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Coronary Arterial Disease (CAD); Surgery (Cardiac); Emotional Freedom Technique
Keywords: coroner arter bypass greft; pain; pain beliefs; anxiety; emotional freedom technique
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Emotional Freedom Technique
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): routine care
- Experimental group (Experimental): Emotional freedom technique
  Interventions: Behavioral: emotional freedom technıque

INTERVENTIONS:
Behavioral: emotional freedom technıque — EFT application
  Other Names: EFT
  Arms: Experimental group

SUMMARY:
When the literature is examined, there is almost no application of EFT on surgical patients. In a quasi-experimental study conducted by Kalroozi et al. (2022) with 70 women who underwent breast cancer surgery and received complementary treatment, the effect of EFT on sleep quality and happiness level was investigated. Six sessions of EFT were applied to the control group. A statistically significant difference was found between the intervention and control groups in sleep quality and happiness scores before and after the intervention. In a randomised controlled study conducted by Menevşe et al. (2024) examining the effect of EFT applied to patients before laparoscopic cholecystectomy on surgical fear and anxiety, 56 patients were included in the control and 56 patients in the intervention group. While routine care and treatment practices were applied to the control group, EFT was applied to the intervention group. EFT application was continued for three rounds and approximately 25-30 minutes. As a result of the study, it was found that EFT was useful in clinical practice in the preoperative period and reduced surgical anxiety and surgical fear. In a quasi-experimental study involving 108 people in which the effects of EFT and music on anxiety and vital signs were examined before lumbar disc herniation surgery, it was found that both music and EFT reduced anxiety and regulated vital signs before surgery, and EFT was more effective than music in regulating anxiety and respiratory rate. In previous studies, pain, pain belief and anxiety in surgical patients have not been examined together. It is thought that the study will have a positive effect on the patient outcomes (anxiety, pain, pain belief) of patients undergoing CABG, thus increasing the holistic approach in the care of patients and having a positive effect on the quality of life of individuals.

DETAILED DESCRIPTION:
Cardiovascular diseases are among the most important causes of mortality and morbidity rates occurring in the world and in our country every year despite the developing technology and treatment methods (1).When the Death and Cause of Death statistics of the Turkish Statistical Institute for 2023 are examined, it is seen that the mortality rate due to circulatory system diseases is 33.4% (2).In the treatment of heart diseases, surgical treatment is frequently preferred in addition to medical treatment. The most commonly used surgical method is open heart surgery (1).Coronary Artery Bypass Graft (CABG) surgery provides re-blooding, oxygenation and nutrition of the non-blooded heart tissue by using artery or vein between the aorta in cases of stenosis or occlusion in the structure of the coronary vessels. CABG is a frequently used method in the world and in our country (3). Regardless of the source of surgical intervention, it causes anxiety in patients. When the literature is examined, it is seen that anxiety is experienced in the majority of surgical patients (4). Fear of death and the unknown, complications that may develop after surgery, pain, loss of organ and independence are among the main causes of anxiety (4). In a study in which anxiety levels of patients who will undergo open heart surgery were examined, preoperative anxiety level was found to be 55.80% (5).The vital importance of the heart increases the fear of death and forms the basis of anxiety in the preoperative and postoperative period (1). In the review, it was found that there were descriptive studies on preoperative anxiety of CABG patients (6, 7, 8, 9), and intervention studies were mostly performed in the form of scent sniffing (10), acupressure (11) music therapy (12,13,14) education (13,15,16); emotional freedom technique was not used.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* No infections, sores in the touch areas
* No psychiatric medication
* No hearing and vision problems
* Stable vital parameters

Exclusion Criteria:

* Patients undergoing re-operation
* Postoperative complications (bleeding, delirium, arrhythmia, etc.)
* Reintubation after extubation
* Drug and stimulant users
* Sedated for more than 24 hours
* Patients unstable for more than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
VAS scale | Pre-test before surgery; post-test 24-48 hours after surgery
  Pain
Pain Belief Scale | Pre-test before surgery; post-test 24-48 hours after surgery
  Pain belief
State Anxiety Scale | Pre-test before surgery; post-test 24-48 hours after surgery
  Anxiety

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ondokuz Mayıs Unıversity, Samsun, Atakum
  - Samsun Training and Research Hospital, Samsun, İlkadım

IPD SHARING:
Plan to Share IPD: Undecided
This is a master thesis. sharing can be done at the end of the study